CLINICAL TRIAL: NCT06928324
Title: Providing Postoperative Analgesia With an Erector Spinae Plane Block in Robotic-assisted Partial Nephrectomy
Brief Title: Postoperative Analgesia With an Erector Spinae Plane Block in Robotic-assisted Partial Nephrectomy
Acronym: ESBPblock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kudret Dogru, Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/114
Record Dates: First submitted 2025-03-24; First posted 2025-04-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Analgesia
Keywords: pain, prostatectomy; erector spinae block
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Active Comparator): Receiving ESPB 30 ml bupivacaine 0.25%
  Interventions: Procedure: Erector Spinae Plane block
- control group (Active Comparator): Not receiving ESBP
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Erector Spinae Plane block — The Erector Spinae Plane Block (ESPB) is a technically simple and safe form of regional anesthesia that can provide effective analgesia for 12 hours in patients with acute postoperative pain
  Other Names: ESBP Block
  Arms: ESPB group
Procedure: Control — No intervention
  Other Names: Not ESBP Block
  Arms: control group

SUMMARY:
Partial nephrectomy is used as a standard method for the treatment of T1 kidney tumors, while radical nephrectomy is preferred for T2 tumors and localized masses that cannot be treated with partial nephrectomy. These surgical procedures can be performed using open surgery, laparoscopic, or robotic approaches. Open surgical methods, especially during partial or radical nephrectomy, generally require wide incisions extending below the costal arch. These incisions involve cutting through intercostal muscle structures, fascial layers, and subcutaneous tissues, which can lead to significant postoperative discomfort for the patient. This situation can directly affect the patient's comfort and recovery time. This study aims to investigate the effect of the erector spinae plane block, a method we routinely use for analgesic purposes in many procedures in anesthesia practice, on postoperative pain levels, analgesic consumption, patient satisfaction, and length of stay after robotic-assisted partial nephrectomy surgery.

Method: Patients ranging in age between 18 and 70 were randomly assigned to either Group 1 (ESPB 30 ml bupivacaine 0.25%) or Group 2 (Control)

DETAILED DESCRIPTION:
Ultrasound-guided regional anesthesia techniques stand out as an effective analgesia method in patients undergoing robotic-assisted partial nephrectomy (RAPN). In recent years, one of the newly defined plane blocks under ultrasound guidance, the Erector Spina Plane (ESP) Block, has become a notable alternative in postoperative pain management (4-6). The ESP block is applied at the level of the spinous process of the T8 vertebra, providing a wide sensory block in the dermatomes from T5 to T12. This technique is performed intraoperatively when the patients are in the lateral decubitus position under general anesthesia, using an ultrasound-guided linear probe. In this study, the effects of the ESP block applied to provide intraoperative and postoperative analgesia in patients undergoing robotic-assisted partial nephrectomy on postoperative pain control will be evaluated. The effectiveness of the ESP block will be comprehensively analyzed in terms of parameters such as reducing pain levels, decreasing analgesic use, increasing patient comfort, and accelerating the postoperative recovery process. Within the scope of this prospective study, general anesthesia induction will be performed using propofol and rocuronium by standard protocols, and anesthesia maintenance will be achieved with a 4-6% combination of desflurane-O₂, remifentanil, and rocuronium intravenous infusion. All procedures will be conducted within an observational clinical research protocol framework, and patients will not be subjected to any methods other than routine practices. Before the study begins, patients will be thoroughly informed, and their written consent will be obtained. The study is planned to start in April 2025.

The patient groups that will not be included in the study are as follows:

* Patients classified as ASA III or IV,
* Patients with cardiopulmonary difficulties,
* Patients who have previously been diagnosed with diabetes,
* Conditions requiring emergency surgery,
* Patients who refuse to participate in the study,
* Individuals with contraindications for general anesthesia,
* Patients with less than 50 kg or more than 110 kg. Patients will be placed in the lateral decubitus position during the surgical procedure, and the surgical site will be prepared under sterile conditions. The Erector Spina Plan (ESP) block will be performed under ultrasound guidance as usual, using a Stimuplex block needle (30-degree angled, 21Gx4", 0.80x100) for this purpose. The block procedure will be performed at the level of the transverse process of the T8 vertebra. Throughout the surgical procedure, vital parameters (systolic, diastolic, and mean arterial pressure, heart rate, and SpO₂) will be regularly recorded at five-minute intervals. The amount of remifentanil used according to analgesic requirements will be systematically recorded during the intraoperative period. The patients' pain levels and analgesic needs will be assessed in the postoperative period at 1, 12, and 24 hours. In addition, the amount of morphine consumed and the need for additional analgesics based on postoperative analgesia requirements will be recorded in detail in both groups. Postoperative pain management will be provided using a patient-controlled analgesia (PCA) device by routine protocols. The PCA device offers effective and reliable pain control by allowing patients to meet their analgesic needs on an individual level. Patients will undergo robotic-assisted partial nephrectomy, and by the surgical procedure, postoperative pain management will be monitored for 24 hours, with potential complications being meticulously recorded. Postoperative pain levels will be assessed in patients both at rest and during coughing using a 0-10 Visual Analog Scale (VAS). When the pain score exceeds 3/10, 1000 mg of intravenous paracetamol will be administered as a rescue analgesic. The time of the patients' first mobilization will be recorded, and the satisfaction level of both the surgeon and the patient during the postoperative period will be rated as 1 (Excellent), 2 (Good), and 3 (Poor). Additionally, the presence of side effects such as nausea and vomiting will also be carefully recorded. Before the study, a power analysis was conducted within the framework of the central hypothesis, based on the postoperative pain rates in both groups, using the G Power (3.1.9.7 Franz Faul, Universität Kiel, Germany) program. According to data obtained from retrospective studies (6), the average morphine consumption in the group where the ESP block was applied was determined to be 16 mg. Based on the assumption that a 30% difference is clinically significant according to the unpaired t-test, a minimum of 38 patients is required for each group. However, 46 patients will be included to increase the evidence for the study.

With this calculation, the power of the study has been determined to be 0.95 and the significance level (α) to be 0.05. The normality of the data will be evaluated using the Shapiro-Wilk test, and homogeneity will be assessed using the Levene test. For data showing a normal distribution, an independent t-test will be used; for data that do not follow a normal distribution or are not homogeneous, the Mann-Whitney U test will be used; and for categorical variables, the Chi-square test will be used. The statistical significance level will be accepted as p<0.05, and all analyses will be conducted using the Windows-compatible JAMOVI (version 2.6.19) software.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I or II
* Having regular preoperative visits
* Pregnant aged 18-70

Exclusion Criteria:

* Patients classified as ASA III or IV,
* Patients with cardiopulmonary difficulties,
* Patients who have previously been diagnosed with diabetes,
* Conditions requiring emergency surgery,
* Patients who refuse to participate in the study,
* Individuals with contraindications for general anesthesia,
* Patients who weighed less than 50 kg or more than 110 kg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Reducing patient-controlled analgesic consumption | From the patient's anesthesia induction in the operating room to the postoperative 24. hours
  The amount of analgesic consumption first 24 hours in the postoperative period

SECONDARY OUTCOMES:
the satisfaction of the surgeon and the patient during the postoperative period | From the patient's anesthesia ending to the postoperative 24. hours
  1 (Excellent), 2 (Good), and 3 (Poor)

CONTACTS AND LOCATIONS:
Overall Officials: Kudret Doğru, Study Director — TC Erciyes University
Locations (1):
- Kudret Doğru, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No